CLINICAL TRIAL: NCT04923685
Title: MicroRNA Correlates of Childhood Maltreatment and Suicidality
Status: Recruiting | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Yogesh Dwivedi, PhD, Professor, University of Alabama at Birmingham
Other Study IDs: IRB-300006024; 5R01MH124248-02 (NIH)
Record Dates: First submitted 2021-06-02; First posted 2021-06-11 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Major Depressive Disorder; Suicidal Ideation
Keywords: Depression; Suicidal Ideation; Suicidality; Healthy Control; Depression and Anxiety; Childhood Maltreatment
MeSH Terms: conditions — Depressive Disorder, Major; Suicidal Ideation; Depression; Anxiety Disorders | interventions — Psychological Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood and urine collection
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (6):
- MDD with elevated CM and suicidality scores: Major Depressive Disorder with elevator childhood maltreatment and suicidality scores.
  Interventions: Other: Trier Social Stress Test
- MDD with CM history but lower suicidality: Major Depressive disorder with childhood maltreatment history but lower suicidality scores.
  Interventions: Other: Trier Social Stress Test
- MDD without CM but with elevated suicidality: Major Depressive Disorder without childhood maltreatment, but with elevated suicidality scores.
  Interventions: Other: Trier Social Stress Test
- MDD without CM but with lower suicidality: Major Depressive Disorder without childhood maltreatment but with lower suicidality scores.
  Interventions: Other: Trier Social Stress Test
- Healthy controls with CM history: Healthy controls with childhood maltreatment history,
  Interventions: Other: Trier Social Stress Test
- Healthy controls without CM history: Healthy controls without childhood maltreatment history.
  Interventions: Other: Trier Social Stress Test

INTERVENTIONS:
Other: Trier Social Stress Test — The TSST is a standardized test to induce acute psychological stress in humans. Participants will abstain from caffeine for 12 hours and nicotine for 2 hours prior to the test. An IV butterfly catheter will be placed in an arm vein and flushed with saline. Participants will rest for 15 minutes. A 10ml baseline blood sample will be drawn. They will perform the TSST task and then have 10ml of blood drawn at 0, 15, 30, 60, and 90 minutes post-TSST.
  Other Names: TSST

SUMMARY:
This is a research study to find out if childhood trauma and stress are associated with depression or suicidal risk. The study will assess the effects of both short-term and long-term stress on biomarker (e.g. miRNA [MiRNA]) levels. miRNAs are a type of RNA (genetic material that is translated into protein) that are found in throughout the body and blood. They are called microRNA because their size is much smaller than typical RNA molecules. miRNAs are highly responsive to environment. This responsiveness is reflected in their expression in individuals who are affected by environment such as stress. The investigators are gathering genetic material, including DNA and RNA, from each participant. The RNA will be taken from the small vesicles and cells in the participant's blood and analyzed. The vesicles are small objects that occur normally in the blood and that contain RNA. This information may help us to understand the cause of mental illness and to improve medical and psychiatric care in the future. There will be 450 participants enrolled in this study.

DETAILED DESCRIPTION:
The purpose of the study is to determine if the relationship between a history of childhood maltreatment (CM) and suicide risk is associated with alterations in the expression and epigenetic modification of specific microRNAs (miRNAs), thereby providing a molecular signature of suicide risk in people with CM. miRNAs are short regulatory RNAs that transduce environmental events into changes in protein synthesis in cells. The environment can induce permanent changes in miRNA expression. Aim 1 is to identify a set of neural-derived exosomal miRNAs that are associated with the interaction of suicidality and CM. Aim 2 is to examine whether an acute experimental stressor, the Trier Social Stress Test (TSST), impacts the expression of these miRNAs in suicidal patients with and without CM. Aim 3 will examine potential mechanisms by which altered miRNAs may contribute to CM-associated suicidal behavior. Aim 4 will examine if changes in CM-associated miRNAs are explained by modifications in their DNA methylation.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-60
2. Physically healthy
3. Willing and able to provide informed consent

5. Diagnosis of MDD or No history of mental illness

Exclusion Criteria:

1. Pregnancy or lactation (women of reproductive potential must have a negative urine pregnancy screen)
2. Post-partum state (being within 2 months of delivery or miscarriage)
3. Homicide risk as determined by clinical interview
4. A lifetime history of psychotic disorder
5. Any history of dissociation or dissociative disorder
6. Bipolar disorder
7. Pervasive developmental disorder
8. Cognitive disorder
9. Cluster A personality disorder
10. Borderline personality disorder
11. Anorexia nervosa
12. Alcohol or drug dependence (except nicotine and caffeine) within the last month or the use of any hallucinogen (except cannabis), including phencyclidine in the last month (NOTE that a positive UDS is not exclusionary except for hallucinogens, methamphetamine, or cocaine. People presenting intoxicated with alcohol may be included when a Breathalyzer test (Alco-Sensor IV) is negative as long as there is no history of recent dependence.
13. Recent myocardial infarction
14. Unstable angina
15. Active neoplasm in the past 6 months
16. Immunosuppressive or corticosteroid therapy within the last month, with the following exceptions: any inhaled, intranasal, topical or vaginal corticosteroids are allowed.
17. Chemotherapy
18. Head injury with loss of consciousness in the past 6 months

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: People between the ages of 18 and 60 with either a history of Major Depressive Disorder or no lifetime history of any major mental illness.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2021-02-26 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
MicroRNA response to stress | 24 hours
  MiRNAs methylation levels will be examined

CONTACTS AND LOCATIONS:
Overall Officials: Yogesh Dwivedi, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (2):
- United States (2):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - UAB Huntsville Regional Medical Campus, Huntsville, Alabama